CLINICAL TRIAL: NCT02924337
Title: A Randomised, Double-blind, Placebo and Active Controlled Crossover Study to Assess the Effect of Single Dose Administration of 2 Doses of Imeglimin on QT/QTc Intervals in Healthy Subjects
Brief Title: Effect of Imeglimin on QT/QTc Intervals in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PXL008-016; 2016-001821-14 (EudraCT Number)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Qt Interval, Variation in
Keywords: QT/QTC interval; Hypoglycemic Agents; Imeglimin; Healthy Volunteers
MeSH Terms: interventions — imeglimin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Imeglimin therapeutic dose (Experimental): Tablet, oral, single dose
  Interventions: Drug: Imeglimin
- Imeglimin supratherapeutic dose (Experimental): Tablet, oral, single dose
  Interventions: Drug: Imeglimin
- Placebo (Placebo Comparator): Tablet, oral, single dose
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Tablet, oral, single dose (400 mg)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Imeglimin
  Arms: Imeglimin supratherapeutic dose; Imeglimin therapeutic dose
Drug: Moxifloxacin
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to assess the effect of a single therapeutic dose and a single supra-therapeutic dose of imeglimin on the QT/QTc interval

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* BMI between 18.5 and 29.9 kg/m2
* weighing between 55 and 95 kg
* willing to use reliable contraception
* able to give fully informed written consent.

Exclusion Criteria:

* Pregnant or lactating woman, or sexually active woman of child-bearing potential not using highly effective contraception
* clinically relevant abnormal medical history, surgery or concurrent medical condition; acute or chronic illness
* clinically significant QT/QTc interval prolongation at Baseline
* history of drug-induced or risk factors for Torsade de Pointes
* any contraindication to moxifloxacin
* severe adverse reaction to any drug or sensitivity to the trial medication or its components
* significant food allergy; use of vitamins, herbal medicines, prescription or over-the-counter medication (with the exception of paracetamol [acetaminophen] and oral contraceptives for women) within 20 days or 6 half-lives before first dose of trial medication
* participation in other clinical trials of unlicensed or prescription medicines, or loss of more than 400 mL blood, within the 3 months before first dose of trial medication
* drug or alcohol abuse; smoking of more than 5 cigarettes, 1 cigars or 1 pipes daily
* regular consumption of more than 5 cups of caffeinated drinks per day
* positive test for hepatitis A, B & C, HIV
* objection by a General Practitioner.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF (deltaQTcF) | Up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Julie Dubourg, MD, Study Director — Poxel SA; Pascale Fouqueray, MD, PhD, Study Director — Poxel SA
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom

REFERENCES:
- [Derived] Dubourg J, Perrimond-Dauchy S, Felices M, Bolze S, Voiriot P, Fouqueray P. Absence of QTc prolongation in a thorough QT study with imeglimin, a first in class oral agent for type 2 diabetes mellitus. Eur J Clin Pharmacol. 2020 Oct;76(10):1393-1400. doi: 10.1007/s00228-020-02929-6. Epub 2020 Jun 18. PMID 32556539